CLINICAL TRIAL: NCT03026023
Title: A Proof of Concept Study for Preemptive Treatment With Grazoprevir and Elbasvir in Donor HCV-positive to Recipient HCV-negative Cardiac Transplant
Brief Title: Preemptive Zepatier Treatment in Donor HCV Positive to Recipient HCV Negative Cardiac Transplant
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: moved forward with another protocol utilizing pan genotypic treatment once it became commercially available and FDA approved
Sponsor: Raymond T. Chung, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Raymond T. Chung, MD, Director of Hepatology, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017P000074
Record Dates: First submitted 2017-01-13; First posted 2017-01-20 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Cardiac Transplant Disorder; Hepatitis C
Keywords: Heart Transplant; Cardiac Transplant; Hepatitis C; Zepatier
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir; elbasvir; elbasvir-grazoprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with grazoprevir + elbasvir +/- ribavirin (Experimental): 12 to 16 weeks of treatment with combination tablet of grazoprevir + elbasvir +/- ribavirin
  Interventions: Drug: Combindation treatment with Grazoprevir and Elbasvir fixed dose combination tablet, with or without ribavirin

INTERVENTIONS:
Drug: Combindation treatment with Grazoprevir and Elbasvir fixed dose combination tablet, with or without ribavirin — HCV treatment for 12 to 16 weeks. Treatment length and addition of ribavirin based upon presence of baseline resistance associated variant in the HCV virus. Medications given concurrently.
  Other Names: Zepatier

SUMMARY:
This is a proof of concept, single center study for the donation of HCV-positive hearts to HCV negative recipient patients, with preemptive, interventional treatment with 12-16 weeks of grazoprevir and elbasvir (with or without ribavirin) to prevent HCV transmission upon transplantation.

DETAILED DESCRIPTION:
Phase 1 of this study will be a single case study with only one subject enrolled. Once safety has been demonstrated and HCV infection transmission shown to be prevented by the protocol, the study will expand to 10 additional patients.

Patients will be selected based on their diminished likelihood of receiving a heart from the waitlist within a period during which they would be likely to succumb to severe comorbidities. This will be determined in part through use of a patient's listing status (1A, 1B, 2) and clinical judgment, and the Seattle Heart Failure Model.

ELIGIBILITY:
Inclusion Criteria:

* Recipient is Age ≥ 18 years
* Serum ALT within normal limits with no history of liver disease
* Lack of sensitization (i.e. PRA < 20%) that would be expected to result in a high likelihood of needing aggressive immunosuppression to treat rejection

Exclusion Criteria:

* Sensitization (i.e. PRA >20%)
* Any liver disease in recipient
* Albumin < 3g/dl or platelet count < 75 x 103/mL
* Need for dual organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Undetectable HCV | 12 Weeks post treatment
  Negative HCV viral RNA at 12 weeks after the last dose of treatment.

SECONDARY OUTCOMES:
Safety and tolerability (based on number of adverse events and out of range lab values) of grazoprevir and elbasvir (with or without ribavirin) in patients who have undergone cardiac transplantation | Upto 16 Weeks
  Safety and tolerability of grazoprevir and elbasvir in the cardiac transplant patient will be monitored by quantifying the number of treatment related adverse events per patient and evaluating out of range laboratory results as compared to baseline/pretreatment values per patient.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond T Chung, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Masschusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified patient data will be shared with research collaborators for safety and data analysis.